CLINICAL TRIAL: NCT06619938
Title: Effects of Using a Consumer-Grade Wearable Device with Biofeedback and Brief Mindfulness Training for Stress Reduction in Family Caregivers of People with Dementia: a Randomized Controlled Trial
Brief Title: Mindfulness-Based Intervention Using Consumer-Grade Wearable Devices with Biofeedback for Family Caregivers of People with Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBA20240927
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Caregiving Stress
MeSH Terms: conditions — Caregiver Burden | interventions — Mindfulness; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Without Biofeedback (Active Comparator)
  Interventions: Behavioral: Mindfulness Without Biofeedback
- Mindfulness With Biofeedback (Experimental)
  Interventions: Behavioral: Mindfulness With Biofeedback

INTERVENTIONS:
Behavioral: Mindfulness With Biofeedback — The intervention includes two weekly 90-minute sessions of brief mindfulness training, covering mindfulness practices, psychoeducation on caregiving, and group sharing. After the first session, participants receive a wearable device for biofeedback on RR, HR, HRV, EDA, and sleep patterns to support mindfulness practice and reduce stress. A 30-minute session teaches caregivers how to use the devices and understand the parameters. The study uses Fitbit Sense with Fitbit apps, employing PPG sensors. The Fitbit Sense connects to smartphones with the apps installed. Caregivers can: (1) view real-time RR, HR, HRV, and EDA on the device and trends on their phone; (2) receive mindfulness practice reminders; (3) access audio coaching; (4) set personal goals (e.g., 30 minutes of daily practice); (5) track practice duration; (6) rate daily stress; and (7) review sleep quality. After the second session, caregivers practice mindfulness for 30 minutes daily over eight weeks.
  Arms: Mindfulness With Biofeedback
Behavioral: Mindfulness Without Biofeedback — The control group will receive two weekly sessions of brief mindfulness training, the same as the intervention group. After the 1st brief mindfulness training, the control group will receive a 30-minute briefing session on goal setting for mindfulness practice. Each caregiver will be asked to develop an action plan for continuous mindfulness practice. A mindfulness therapist will also discuss the challenges and solutions for developing a habit of mindfulness practice with the caregivers in the second session. Caregivers in the control group will be advised to practice mindfulness daily for 30 minutes over the course of eight weeks.
  Arms: Mindfulness Without Biofeedback

SUMMARY:
The aim of this study is to investigate the effectiveness of a brief mindfulness training intervention using a consumer-grade wearable device with biofeedback for reducing stress and promoting psychological health in family caregivers of people with dementia.

The intervention includes two weekly sessions, each lasting 90 minutes, of brief mindfulness training. The intervention group will be provided with a wearable device that offers biofeedback, which aims to promote their mindfulness practice and help the caregivers cultivate a mindful attitude in their daily activities, leading to stress reduction. Participants in the intervention group will attend a 30-minute briefing session to learn how to use the wearable device and understand the parameters displayed on the device. The caregivers will be instructed to practice mindfulness for 30 minutes every day over the course of eight weeks.

Participants will be randomly assigned to receive either the mindfulness intervention combined with biofeedback or the mindfulness intervention alone. Evaluations will be conducted at three time-points: baseline (0 weeks), mid-intervention (4 weeks), and post-intervention (8 weeks). Both groups will complete the same assessments at each time-point.

DETAILED DESCRIPTION:
Family caregivers of people with dementia (PWD) face significant challenges in managing various caregiving tasks and addressing behavioral issues exhibited by their care recipients. The burden of caregiving and uncertainty about disease progression can lead to high levels of stress among these caregivers. Providing community resources and support for PWD caregivers, particularly to reduce caregiving stress, is crucial and highly recommended. Mindfulness training has been identified as an effective intervention for stress reduction in PWD caregivers. However, maintaining a regular mindfulness practice is essential for achieving sustainable stress reduction, and long-term adherence to self-practice remains a challenge for family caregivers. To help maintain their mindfulness practice, providing participants with visualized improvement via biofeedback may be beneficial.

Biofeedback, a self-regulation technique that helps individuals voluntarily control their automatic body functions, has shown promise in stress reduction. By measuring physiological parameters such as respiratory rate (RR), heart rate (HR), heart rate variability (HRV), and electrodermal activity (EDA), individuals can gain greater awareness of their body's functioning and recognize health problems, motivating them to modify their lifestyle and reduce stress. Previous studies on biofeedback training have primarily been conducted in laboratory or clinical settings, requiring the presence of a therapist and using large, expensive medical monitors. However, the recent proliferation of consumer-grade wearable devices, such as the Apple Watch and Fitbit, offers a more accessible, affordable, and user-friendly alternative. These devices provide self-directed learning and biofeedback, including RR, HR, HRV, EDA, and sleep patterns. Unlike medical-grade monitors, consumer-grade wearables often present health parameters in simple figures and graphics, making it easier for users to understand their stress levels. Moreover, validation studies have demonstrated high agreement between consumer-grade and medical-grade devices for various parameters in diverse populations, including patients with chronic obstructive pulmonary disease, pediatric patients, intensive care unit patients, and cardiac rehabilitation patients. Additionally, these lightweight, waterproof devices can continuously measure and provide information about daily stress patterns, activities, and the effects of relaxation skills and mindfulness practice.

This study aims to investigate the effectiveness of a brief mindfulness-based intervention combined with biofeedback using consumer-grade wearable devices in reducing stress among family caregivers of PWD. The study will also examine secondary outcomes, including heart rate variability, depressive symptoms, anxiety symptoms, trait mindfulness, and neuropsychiatric symptoms in care recipients.

The target population for this study will be family caregivers of PWD. They will be recruited from elderly centers through collaborations with local non-governmental organizations. Interested participants will be assessed for eligibility. After interested and eligible participants provide their consent, they will be randomly assigned to receive either the mindfulness intervention combined with biofeedback or the mindfulness intervention alone.

The intervention includes two weekly sessions (90 minutes each) of brief mindfulness training. After the first session of mindfulness training, the intervention group will be given a wearable device with biofeedback on RR, HR, HRV, EDA, and sleeping patterns, which aims to promote their mindfulness practice and help the caregivers cultivate a mindful attitude in their daily activities, leading to stress reduction. A 30-minute briefing session will be provided for the caregivers to learn how to use the wearable devices and understand the parameters on the device. In this study, the Fitbit Sense with the Fitbit apps will be used. The caregivers can (1) receive real-time RR, HR, HRV, and EDA on the wearable device and review the trends on their smartphone; (2) receive a daily reminder for mindfulness practice from the wearable device; (3) listen to audio coaching for mindfulness practice from the Fitbit apps; (4) set a personal goal (e.g., daily practice of 30 minutes) in the Fitbit apps; (5) track and record their duration of practice; (6) rate and review their perceived daily stress level; and (7) review their duration and quality of sleep. After the second session of brief mindfulness training, the caregivers will be instructed to practice mindfulness for 30 minutes every day over the course of eight weeks.

The control group will receive two weekly sessions of brief mindfulness training, the same as the intervention group. After the first brief mindfulness training, the control group will receive a 30-minute briefing session on goal setting for mindfulness practice. Each caregiver will be asked to develop an action plan for continuous mindfulness practice. A mindfulness therapist will also discuss the challenges and solutions for developing a habit of mindfulness practice with the caregivers in the second session. All caregivers in both the intervention and control groups will be advised to practice mindfulness daily for 30 minutes.

The outcome measures assessed include perceived caregiving stress (primary), heart rate variability, depressive symptoms, anxiety symptoms, trait mindfulness, and neuropsychiatric symptoms. Feasibility measures include eligibility and enrollment, attendance rate, adherence rate, and retention rate. Evaluations will be conducted at baseline (0 weeks), mid-intervention (4 weeks), and post-intervention (8 weeks). Both groups will complete the same assessments at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of an individual who has been residing in the community with a confirmed medical diagnosis of any type of dementia (from NGO record or the care-recipients' medical record);
* Providing care for at least 4 hours or more per week;
* Able to speak Cantonese (for understanding all teaching materials and instructions).

Exclusion Criteria:

* Practicing or having recently learned meditation, mindfulness activities, and/or relaxation training in the last 6 months;
* Regularly using wearable devices;
* Diagnosed with a mental disorder such as bipolar disorder, schizophrenia, dementia, or depression in an acute phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Perceived Caregiving Stress in the Family Caregiver | 8 Weeks
  The Perceived Stress Scale (PSS) comprises 10 items rated on a 5-point Likert Scale (0 = never to 4 = very often) to assess perceived stress levels. The total score varies from 0 to 40, with a higher score reflecting more perceived stress. Scores within the ranges of 0-13, 14-26, and 27-40 correspond to low, moderate, and high levels of perceived stress, respectively.

SECONDARY OUTCOMES:
Depressive Symptoms in the Family Caregiver | 8 Weeks
  The Center for Epidemiologic Studies Depression Scale (CESD) comprises 20 items rated on a 4-point Likert scale (0 = rarely or none of the time to 3 = most or almost all the time) to assess the severity of depressive symptoms experienced in the past week. The total score ranges from 0 to 60, with a higher score indicating more severe depressive symptoms. Scores within the ranges of 0-14, 15-21, and 22-60 correspond to low, mild to moderate, and a potential indication of major depression, respectively.
Heart Rate Variability (HRV) in the Family Caregiver | 8 Weeks
  HRV will be measured as a biomarker of stress. The interpretation of HRV will follow the Guidelines for Standard Measurement and Interpretation of HRV (European Society of Cardiology and the North American Society of Pacing and Electrophysiology) using the frequency-domain method.
Anxiety in the Family Caregiver | 8 Weeks
  The Hospital Anxiety and Depression Scale-Anxiety (HADS-A) measures generalized anxiety, including tension, worry, fear, panic, difficulties in relaxing, and restlessness. It consists of 7 items and is rated on a 4-point Likert scale. A higher score on the HADS-A suggests a higher level of anxiety.
Trait Mindfulness in the Family Caregiver | 8 Weeks
  The Five-Facet Mindfulness Questionnaire-Short Form measures trait mindfulness. It consists of 20 items that assess five domains of mindfulness: observing, describing, acting with awareness, nonjudging, and nonreacting. Each domain comprises 4 items and is rated on a 5-point Likert scale (1 = never, 5 = very often). The facet score for each domain is the average of the four items, with higher scores (range = 1-5) indicating higher levels of mindfulness.
Neuropsychiatric Syndromes in the Care Recipient | 8 Weeks
  The Neuropsychiatric Inventory (NPI) measures neuropsychiatric syndromes that occur in Alzheimer's disease and other neurodegenerative disorders. The NPI is administered by the family caregiver and consists of the following domains: Delusions, Hallucinations, Agitation/Aggression, Depression/Dysphoria, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability/Lability, and Aberrant Motor Behavior. Each domain is rated based on its frequency (1 = rarely, less than once per week; 4 = very often, once or more per day) and severity (1 = mild, producing little distress in the patient; 3 = severe, very disturbing to the patient and difficult to redirect). A total score can be obtained for each domain by multiplying the frequency and severity ratings. The total score of the NPI is obtained by summing the scores across all domains, with a higher score indicating more severe neuropsychiatric syndromes.
Feasibility of Eligibility and Enrollment | 8 Weeks
  The number of eligible participants and the proportion of those eligible who enrolled will be assessed.
Feasibility of Attendance Rate | 8 Weeks
  The number and proportion of participants who attended will be assessed.
Feasibility of Adherence to Wearing the Wearable Device | 8 Weeks
  Adherence to wearing the wearable device will be measured by the number of times the physiological data is reviewed per day.
Feasibility of Retention Rate | 8 Weeks
  The number and proportion of participants completing all assessments will be assessed.

IPD SHARING:
Plan to Share IPD: No